CLINICAL TRIAL: NCT01406574
Title: A Multicenter, Open-label, Non-randomized, Dose-escalation, Therapeutic Exploratory Trial to Evaluate the Safety and Efficacy of OPB-31121 in Patients With Progressive Hepatocellular Carcinoma
Brief Title: Phase I/II Study of OPB-31121 in Patients With Progressive Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 252-11-001; JapicCTI-111546 (Other: JAPIC)
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OPB-31121 p1 (Experimental): Phase1 step
  Interventions: Drug: OPB-31121
- OPB-31121 p2 (Experimental): Phase2 step
  Interventions: Drug: OPB-31121 phase2

INTERVENTIONS:
Drug: OPB-31121 — Oral administration, 400 mg/day or 600 mg once daily after breakfast during the treatment period (1 month)
  Arms: OPB-31121 p1
Drug: OPB-31121 phase2 — Oral administration, recommended dose from Phase1 once daily after breakfast during the treatment period (6 months)
  Arms: OPB-31121 p2

SUMMARY:
The purpose of this study is:

Phase1: To evaluate the safety and determine the recommended dose (RD) Phase2: To evaluate the efficacy

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologically or clinically confirmed diagnosis of hepatocellular carcinoma
* Patients with Child-Pugh classification A or B
* Patients unresponsive to standard therapy or for whom standard therapy is intolerable, or for whom there is no appropriate therapy
* Patients who are able to take oral medication
* Patients age 20 to 79 years (inclusive) at time of informed consent
* Patients with an ECOG performance status score of 0-2
* Patients have the eligible organ function.

Exclusion Criteria:

* Patients with a primary malignant tumor
* Patients with a history of liver transplant
* Patients with brain metastases
* Patients with a complication of uncontrolled
* Patients with a psychiatric disorder that might cause difficulty in obtaining informed consent or in conducting the trial

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Chiba
  - Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- OPB-31121: 50mg/Day; OPB-31121: 100mg/Day; OPB-31121: 200mg/Day; OPB-31121: 400mg/Day: OPB-31121: 50, 100, 200 and 400 mg/day oral once daily (QD) in a 4 week cycle.
Period: Overall Study
Arm/Group | OPB-31121: 50mg/Day | OPB-31121: 100mg/Day | OPB-31121: 200mg/Day | OPB-31121: 400mg/Day
Started | 7 | 4 | 7 | 5
Completed | 6 | 3 | 6 | 1
Not Completed | 1 | 1 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Definite progression of primary disease | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- OPB-31121: OPB-31121: 50, 100, 200 and 400 mg/day oral once daily (QD) in a 4 week cycle.
Arm/Group | OPB-31121
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 20
Region of Enrollment [Number; unit: participants]
  Japan | 23

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Treatment Emergent Adverse Events
Description: Treatment emergent adverse events observed during outcome measure time frame.
Time Frame: From first study medication to on Day 32 (after repeated 28 days medication from Day 4 to 32)
Population: Safety population No statistical analysis provided for Subjects With Treatment Emergent Adverse Events.
Measure: Number; unit: participants
Arm/Group | OPB-31121
Number analyzed (Participants) | 23
participants | 23

2. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs)
Description: Recommended Dose (RD) of OPB-31121 was defined as the highest dose at which Dose Limited Toxicity (DLT) occurred at an incidence of < 30%.
  DLT was defined as adverse events related to OPB-31121 occurring until Day 32, and 1) Grade 4 neutrophil count decreased persisting for ≧ 8 days, or Grade 3 or 4 febrile neutropenia, or infection with neutrophil count decreased 2) Grade 4 Plt decreased, or Grade 3 Plt decreased persisting for ≧ 8 days 3) Grade 3 or 4 nausea, vomiting, or diarrhoea that occurred despite the use of an anti-emetic or anti-diarrheal agents 4) Grade 3 or more severe AEsa excluding the AEs presented above 1) to 3) 5) AEs requiring interruption of IMP administration for a period of ≧ 8 consecutive days 6) Same AEs causing interruption of IMP administration twice
Time Frame: From first study medication to on Day 32 (after repeated 28 days medication from Day 4 to 32)
Population: DLT evaluated subjects who had achieved ≧75% study drug compliance during a 4-week (28-day) treatment period starting from Day 4.
  No statistical analysis provided for Subjects With DLTs.
Measure: Number; unit: participants
Groups:
- OPB-31121: 50 mg/Day; OPB-31121: 100 mg/Day; OPB-31121: 200 mg/Day; OPB-31121: 400 mg/Day: OPB-31121: 50, 100, 200 and 400 mg/day oral once daily (QD) in a 4 week cycle.
Arm/Group | OPB-31121: 50 mg/Day | OPB-31121: 100 mg/Day | OPB-31121: 200 mg/Day | OPB-31121: 400 mg/Day
Number analyzed (Participants) | 7 | 4 | 7 | 5
participants | 0 | 0 | 1 | 4

3. Secondary Outcome: Best Overall Response
Description: Overall response was evaluated based on the Response Evaluation Criteria in Solid Tumors (RECIST guideline) - mRECIST 1.0.
Time Frame: From first dose of study medication up to 28 weeks
Population: Efficacy population included all treated subjects who had received at least 1 dose of study drug.
  No statistical analysis provided for Best Overall Responders.
Measure: Number; unit: participants
Arm/Group | OPB-31121
Number analyzed (Participants) | 23
participants
  CR or PR | 0
  SD ≧ 8w | 6
  PD | 9
  NE | 8

ADVERSE EVENTS:
Time Frame: From first study medication to end-of-trial examination
Arm/Group | OPB-31121: 50 mg/Day | OPB-31121: 100 mg/Day | OPB-31121: 200 mg/Day | OPB-31121: 400 mg/Day
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4 | 0/7 | 2/5
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4 | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPB-31121: 50 mg/Day (N=7) | OPB-31121: 100 mg/Day (N=4) | OPB-31121: 200 mg/Day (N=7) | OPB-31121: 400 mg/Day (N=5)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — General disorders and administration site conditions
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPB-31121: 50 mg/Day (N=7) | OPB-31121: 100 mg/Day (N=4) | OPB-31121: 200 mg/Day (N=7) | OPB-31121: 400 mg/Day (N=5)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 7 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 7 (7) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 6 (6) | 4 (4)
Fatigue/malaise (Gastrointestinal disorders) | 5 (5) | 1 (1) | 4 (4) | 2 (2) — General disorders and administration site conditions
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No